CLINICAL TRIAL: NCT02997618
Title: The AAA Get Fit Trial: A Pilot Randomised Controlled Trial of Community Based Exercise to Improve Fitness and Reduce Morbidity and Mortality of Patients With Abdominal Aortic Aneurysms
Brief Title: The AAA Get Fit Trial: A Pilot Randomised Controlled Trial of Community Based Exercise in Patients With Abdominal Aortic Aneurysms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Charles McCollum, Professor, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 162347
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): 1. Usual care (control)
  Usual care given to patients on AAA surveillance. This includes six-monthly or annual ultrasound measurements of AAA, attendance to surveillance clinic and written (APPENDIX A) and verbal advice on managing cardiovascular risk. This advice will be based on current widely available NHS patient information15 and consists of the following information with regard to:
  Smoking Exercise Weight Diet
  Interventions: Other: Control
- Community Based Exercise Programme (Experimental): Community based-exercise (in addition to usual care) with the choice of either:
  1. Home-based exercise training Participants choosing to exercise at home will follow the programmes intended for this setting, with each exercise designed to be possible without the need for specialist equipment.
  2. Gym-based exercise training Participants will exercise at their nearest Life Leisure LTD gym, following one of the instructor designed programmes , using a combination of aerobic and resistance equipment, as well as simple floor exercises.
  Duration and Frequency At least 50 minutes of exercise per day on three non-consecutive days of the week for 20 weeks.
  Interventions: Behavioral: Community based exercise programme

INTERVENTIONS:
Behavioral: Community based exercise programme — 20 week community (home or gym based) exercise programme
  Arms: Community Based Exercise Programme
Other: Control — Usual care consisting of advice.
  Arms: Control

SUMMARY:
Rupture of abdominal aortic aneurysms(AAA) causes 12,000 deaths/year in the UK.1 Elective repair to prevent this carries a perioperative mortality of 4.5% for open surgery and 1% for endovascular repair. This risk is associated with poor cardiorespiratory fitness which can be measured using Cardiopulmonary Exercise Testing(CPET) with the CPET variables, peak oxygen uptake(peakVO2)<15ml/kg/min and anaerobic threshold(AT)<10.2ml/kg/min identifying patients at increased risk of early death after AAA repair.3 These variables can therefore be used as surrogate markers for cardiovascular fitness and risk of mortality and morbidity in AAA surgery; optimising these markers should improve fitness and decrease this risk. The optimal duration and type of exercise training for improving peak VO2 and AT in AAA patients is not known. AAA patients are unique as they are motivated to reduce the risk of impending surgery but are afforded the time to improve their fitness as repair may not be needed for months or even years.

The investigators propose a pilot randomised controlled trial to explore the effectiveness of a 20-week community (either home or gym-based) exercise programme to achieve sustained improvements in peak VO2 and AT, as measured by CPET, in AAA patients. Changes in QoL, habitual activity levels and cardiovascular risk will also be assessed. The results will inform a definitive multicentre clinical trial on exercise to improve outcomes in elderly patients with cardiovascular disease and AAA.

ELIGIBILITY:
Inclusion Criteria:

1. Men with an AAA ≥ 3.0 and < 5.0 cm and women with a AAA ≥ 3.0 and < 4.5 cm
2. Aged 60 - 85 years inclusive
3. Willing and able to engage in gym- and/or home-based exercise training and undertake CPET

Exclusion Criteria:

1. Unable or unwilling to undertake CPET or exercise training Patients unwilling will not be able to give informed consent and those who are unable would not be able to be randomised to the intervention study group nor undergo satisfactory testing to obtain our outcome measures.
2. High levels of habitual physical activity (those scoring "high" on the PASE questionnaire) These patients already have a high level of physical activity and therefore it may not be possible to improve their fitness any further which is the primary objective of the study.

   Exclusion criteria 3-10 are all based on medical conditions which would mean either exercise training may be unsafe, they would require further investigation and treatment of that medical condition or are likely to need upcoming intervention for their medical condition which would take priority over any participation in a research study. If any medical conditions are discovered during the study, these patients will be withdrawn from the study and referred to the necessary health professional.
3. Severe liver disease (INR > 2, serum albumin < 3.0g/dL, bilirubin > 50µmol/L)
4. Unstable angina, angina of < 2 month's duration, occurring more than twice daily, angina that is increasing in frequency or precipitated by less exertion, angina at rest
5. Uncontrolled atrial fibrillation (AF) or other arrhythmia: untreated paroxysmal AF
6. Moderate or severe aortic valve stenosis (peak systolic pressure gradient >40mmHg or with an aortic valve area < 1cm2)
7. Class II/III/IV heart failure and/or left ventricular ejection fraction < 25%
8. Pericarditis or myocarditis within last six months
9. Patients with > 2mm ST depression on exercise ECG will not be eligible to take part and will be referred to a cardiologist for further assessment.
10. Diagnosis or treatment for a malignancy over the previous 12 months

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 as measured by CPET | at 20 weeks

SECONDARY OUTCOMES:
Anaerobic Threshold as measured by CPET | at 20 weeks
Biomarkers of Cardiovascular disease risk | at 20 weeks
Other risk factors of Cardiovascular disease risk | at 20 weeks
  Weight, BMI, Waist Circumference and Blood Pressure
Subjective measure of habitual activity levels (PASE questionnaire) | at 20 weeks
Objective measure of habitual activity levels (via Accelerometry) | at 20 weeks
Health-related quality of life | at 20 weeks
Early changes in outcome measures | at 10 weeks
  All outcome measures will also be measured at 10 weeks and compared with other time intervals.
Sustainability of changes in outcome measures | at 30 weeks
  All outcome measures recorded 10 weeks post cessation of exercise at 30 weeks and compared with the other time intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Charles McCollum, MD, FRCS, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: Undecided